CLINICAL TRIAL: NCT05152849
Title: A Randomized, Double-Blind, Placebo-Controlled Pilot Study to Evaluate the Efficacy, Safety, and Tolerability of AXA1125 in Subjects With Fatigue-Predominant Post-Acute Sequelae of SARS-CoV-2 (PASC) Infection
Brief Title: Efficacy, Safety, Tolerability of AXA1125 in Fatigue After COVID-19 Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Axcella Health, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AXA1125-201
Record Dates: First submitted 2021-11-29; First posted 2021-12-10 (Actual); Last update posted 2022-10-20 (Actual); Status verified 2021-11

CONDITIONS: Post-Acute Sequelae of SARS-CoV-2 (PASC) Infection
Keywords: Long COVID; Long-haul COVID; Muscle weakness; COVID; PASC; Fatigue; Amino acids; Bioenergetics; Mitochondrial dysfunction; Phosphocreatine recovery; Exertional fatigue; Phospho magnetic resonance spectroscopy; Skeletal muscle
MeSH Terms: conditions — Infections; Post-Acute COVID-19 Syndrome; Muscle Weakness; Fatigue; Mitochondrial Diseases | interventions — leucine, isoleucine, valine, arginine, glutamine, and N-acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AXA1125 33.9g (Experimental): 33.9 g AXA1125 administered orally BID with or without food
  Interventions: Drug: AXA1125
- Placebo (Placebo Comparator): Matching Placebo administered orally BID with or without food
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AXA1125 — AXA1125 administered BID with or without food
  Arms: AXA1125 33.9g
Drug: Placebo — Matching Placebo administered BID with or without food
  Arms: Placebo

SUMMARY:
This study will compare the effects of AXA1125, an orally active mixture of amino acids, compared to placebo, on improving muscle function (metabolism) following moderate exercise in subjects with fatigue-Predominant Post-Acute Sequelae of SARS-CoV-2 as well as the safety and tolerability of AXA1125. Subjects will take one dose of AXA1125 or a placebo twice daily for 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Willing to participate in the study and provide written informed consent
* Male and female adults aged > 18 years and less than 65 years
* Must have had clinically suspected COVID-19 and a positive antibody test or a documented SARS-CoV-2 infection (a positive reverse transcription polymerase chain reaction test) at least 12 weeks prior to Screening
* Must have fatigue-predominant PASC
* Other than PASC, a subject must be in good health without other significant medical or not well controlled medical or psychiatric conditions

Exclusion Criteria:

* Other than PASC, have an explanation for fatigue
* Other than PASC, a history or presence of an uncontrolled, clinically significant disease
* Medical history that includes of Non-invasive or invasive ventilatory support for COVID 19, Intensive care unit or other high dependency unit admission for COVID-19, Hospitalization for >1 week for COVID-19 without intubation

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2022-06-21 (Actual); Study Completion 2022-06-29 (Actual)

PRIMARY OUTCOMES:
Change from baseline at Week 4 in the phosphocreatine (PCr) recovery rate following moderate exercise, as assessed by 31P-magnetic resonance spectroscopy (MRS) | Baseline to 28 days

SECONDARY OUTCOMES:
Change from baseline in PCr recovery rate as assessed by phosphorus magnetic resonance spectroscopy (31P-MRS) | Baseline to 28 days
Proportion of subjects with improvement in PCr recovery rate | Baseline to 28 days
Change from baseline in serum lactate level after a 6-minute walk test | Baseline to 28 days
Proportion of subjects with serum lactate level ≤3 mmol/L after a 6MWT | Baseline to 28 days
Proportion of subjects with a decrease in venous serum lactate level from baseline after a 6MWT | Baseline to 28 days
Change from baseline in distance traveled during a 6MWT | Baseline to 28 days
Change from baseline in subjects' fatigue score as assessed by Chalder Fatigue Questionnaire (CFQ)-11 | Baseline to14 days
Change from baseline in subjects' fatigue score as assessed by Chalder Fatigue Questionnaire (CFQ)-11 before and after a 6MWT | Baseline to 28 days
Proportion of subjects with an improvement in fatigue score as assessed by CFQ-11 before and after a 6MWT | Baseline to 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Betty Raman, MBBS DPhil FRACP, Principal Investigator — Oxford University Hospitals NHS Trust
Locations (1):
- Oxford University Hospitals NHS Foundation Trust, Oxford, United Kingdom

REFERENCES:
- [Derived] Finnigan LEM, Cassar MP, Koziel MJ, Pradines J, Lamlum H, Azer K, Kirby D, Montgomery H, Neubauer S, Valkovic L, Raman B. Efficacy and tolerability of an endogenous metabolic modulator (AXA1125) in fatigue-predominant long COVID: a single-centre, double-blind, randomised controlled phase 2a pilot study. EClinicalMedicine. 2023 May;59:101946. doi: 10.1016/j.eclinm.2023.101946. Epub 2023 Apr 14. PMID 37223439